CLINICAL TRIAL: NCT06475963
Title: Evaluation of Clinical Outcomes of Scaffold Treatment of Partial Meniscal Injuries of the Knee, an Observational Study.
Brief Title: Evaluation of Clinical Outcomes of Scaffold Treatment of Partial Meniscal Injuries of the Knee
Acronym: STAR-ACT
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: STAR-ACT
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis; Knee Injuries; Meniscus Lesion
MeSH Terms: conditions — Osteoarthritis, Knee; Knee Injuries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients: Patients will be recruited from all subjects treated surgically with scaffolds for partial meniscal defects from January 01, 2009 to December 31, 2019
  Interventions: Other: surveys

INTERVENTIONS:
Other: surveys — telephone survey

SUMMARY:
The study consists of 3 phases (Identification of includable patients, Telephone follow-up evaluation and the collection of study-specific clinical data in medical records of enrolled patients):

* Identification by trained medical personnel of subjects who meet the study's inclusion criteria.
* Once the patient's Informed Consent has been obtained, the study-specific questionnaires will be submitted by telephone.
* Study-specific clinical score data will be collected from the medical records of patients enrolled in the study. These data will be used, together with the data collected during the telephone follow-up, to evaluate the trend in outcomes over time after implantation of this scaffold.

ELIGIBILITY:
Inclusion Criteria:

* Acute irreparable meniscal injuries requiring partial meniscectomy or chronic meniscal tissue loss (traumatic or degenerative) greater than 25%; Intact anterior and posterior meniscal horn respectively;
* Peripheral meniscal rim (1 mm or more) along the entire circumference of the involved meniscus;
* Knee stability or anterior cruciate ligament injury stabilized at the time of surgery;
* Male or female patients between the ages of 18 and 65 years;
* Healthy contralateral knee;
* Normal axial alignment of the knee (mechanical tibio-femoral angle < 3°)
* Patients treated surgically with scaffolds (Actifit) for partial meniscal defects from January 01, 2009 to December 31, 2019

Exclusion Criteria:

* Patients no longer available;
* Concomitant posterior cruciate ligament (PCL) injury;
* Advanced cartilage injuries according to Outerbridge classification (IV);
* Incorrect axial alignment of the lower limb;
* Documented allergy to polyurethane;
* Local or systemic infection;
* History of previous anaphylactoid reaction;
* Systemic administration of corticosteroids or immunosuppressive drugs within 30 days prior to surgery;
* Evidence of osteonecrosis in the involved knee;
* Positive history of rheumatoid arthritis, inflammatory arthritis and autoimmune diseases;
* Neurological disorders or conditions that may affect the rehabilitation protocol;
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from all subjects treated surgically with scaffolds (Actifit) for partial meniscal defects from January 01, 2009 to December 31, 2019
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
International Knee Documentation Committee | baseline (post surgery)
  This is a subjective, knee-specific rating scale that is considered one of the most reliable assessment tools in the evaluation of knee pathology. The questionnaire examines 3 categories: symptoms, sports activity, and knee function. According to this questionnaire, a score between 0 and 100 can be obtained, where a high score is associated with a high level of function and minor pain symptoms. A score of 100 is in fact interpreted as a condition in which there are neither limitations in conducting activities of daily living nor symptoms.
Visual Analogue Scale pain | baseline (post surgery)
  It is a one-dimensional quantitative 11-point numeric pain rating scale; the scale requires the patient to select the number that best describes the intensity of his or her pain, from 0 to 10, at that specific time. 0 means no pain and 10 indicates the worst possible pain.
EuroQoL (quality of life) Current Health Assessment | baseline (post surgery)
  Valuable tool for measuring the quality of life of a patient.
EuroQoL Visual Analogue Scale (EQ-VAS) | baseline (post surgery)
  This is a visual analog scale that has a range of scores from 0 (worst imaginable health condition) to 100 (best imaginable health condition).
Tegner Score | baseline (post surgery)
  It allows the estimation of a subject's motor activity level with a score between 0 and 10, where 0 represents 'inability' and 10 represents 'participation in competitive sports, such as soccer at the national or international level. This score is the one most commonly used to define the motor activity level of patients with knee disorders. In the study, the Tegner Score will be compiled directly by the investigator, through an interview the patient.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | baseline (post surgery)
  It is a pathology-specific questionnaire useful for the assessment of symptoms reported at the knee joint level in patients with osteoarthritis.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Houck DA, Kraeutler MJ, Belk JW, McCarty EC, Bravman JT. Similar clinical outcomes following collagen or polyurethane meniscal scaffold implantation: a systematic review. Knee Surg Sports Traumatol Arthrosc. 2018 Aug;26(8):2259-2269. doi: 10.1007/s00167-018-4838-1. Epub 2018 Jan 16. PMID 29340746
- [Result] Condello V, Dei Giudici L, Perdisa F, Screpis DU, Guerriero M, Filardo G, Zorzi C. Polyurethane scaffold implants for partial meniscus lesions: delayed intervention leads to an inferior outcome. Knee Surg Sports Traumatol Arthrosc. 2021 Jan;29(1):109-116. doi: 10.1007/s00167-019-05760-4. Epub 2019 Oct 25. PMID 31654130
- [Result] Filardo G, Kon E, Perdisa F, Sessa A, Di Martino A, Busacca M, Zaffagnini S, Marcacci M. Polyurethane-based cell-free scaffold for the treatment of painful partial meniscus loss. Knee Surg Sports Traumatol Arthrosc. 2017 Feb;25(2):459-467. doi: 10.1007/s00167-016-4219-6. Epub 2016 Jul 9. PMID 27395355
- [Result] Grassi A, Zaffagnini S, Marcheggiani Muccioli GM, Benzi A, Marcacci M. Clinical outcomes and complications of a collagen meniscus implant: a systematic review. Int Orthop. 2014 Sep;38(9):1945-53. doi: 10.1007/s00264-014-2408-9. Epub 2014 Jun 20. PMID 24947329
- [Result] Zaffagnini S, Giordano G, Vascellari A, Bruni D, Neri MP, Iacono F, Kon E, Presti ML, Marcacci M. Arthroscopic collagen meniscus implant results at 6 to 8 years follow up. Knee Surg Sports Traumatol Arthrosc. 2007 Feb;15(2):175-83. doi: 10.1007/s00167-006-0144-4. Epub 2006 Jul 15. PMID 16845545
- [Result] Zaffagnini S, Marcheggiani Muccioli GM, Bulgheroni P, Bulgheroni E, Grassi A, Bonanzinga T, Kon E, Filardo G, Busacca M, Marcacci M. Arthroscopic collagen meniscus implantation for partial lateral meniscal defects: a 2-year minimum follow-up study. Am J Sports Med. 2012 Oct;40(10):2281-8. doi: 10.1177/0363546512456835. Epub 2012 Aug 20. PMID 22915481